CLINICAL TRIAL: NCT02022579
Title: A Multi-Center Study Evaluating the Utility of Diffusion Weighted Imaging for Detection and Diagnosis of Breast Cancer
Brief Title: DCE-MRI and DWI for Detection and Diagnosis of Breast Cancer
Acronym: ACRIN6702
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: American College of Radiology Imaging Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ACRIN 6702; U01CA080098 (NIH); U01CA079778 (NIH)
Record Dates: First submitted 2013-12-16; First posted 2013-12-30 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Breast Cancer; BIRADS 3; BIRADS 4; BIRADS 5
Keywords: Breast Cancer; Diagnosis; Malignant; Benign; Biopsy
MeSH Terms: conditions — Breast Neoplasms; Disease | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DCE-MRI and DWI (Experimental): Single arm study, diagnosis defined as BIRADS 3, 4, or 5 lesion(s) based on DCE-MRI only with DWI collected in tandem as standard practice.
  Interventions: Procedure: DCE-MRI and DWI

INTERVENTIONS:
Procedure: DCE-MRI and DWI — DCE-MRI defined lesion(s) compared with biopsy results or 1-year follow up
  Other Names: magnetic resonance imaging; MRI; DCE-MRI; DWI; DW-MRI

SUMMARY:
A type of magnetic resonance imaging called diffusion weighted imaging (DWI) will be tested to define cancerous from non-cancerous lesions in the breast.

DETAILED DESCRIPTION:
For this study, the investigators plan to evaluate DWI scans performed in women with breast lesions identified by conventional breast MRI. The investigators will determine whether an ADC threshold can be defined for distinguishing benign and malignant lesions on DWI, assess the difference in ADC cutoffs for mass and non-mass lesions, and investigate the potential improvement in accuracy using techniques such as nonzero minimum b-value (to remove perfusion effects in the ADC measures) and normalized ADC measures (to account for variations in water content and other factors).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent;
* 18 years of age or older;
* Successful completion of breast MR examination with DWI required by protocol;
* Undiagnosed breast lesion (BI-RADS 3, 4, or 5) identified on MRI. The BI-RADS assessment must refer to a focal finding within the breast (i.e. mass, non-mass, or focus) as opposed to diffuse processes (e.g. background parenchymal enhancement, skin thickening) or lesions outside the subcutaneous breast (e.g. axillary lymph nodes, focal skin lesions, osseous lesions, etc.).

Exclusion Criteria:

* Participants with current or recent history (within 6 months prior to the MRI) of chemotherapy for cancer;
* Neoadjuvant chemotherapy between MRI and confirmation of lesion outcome (study lesions must be biopsied prior to undergoing any chemotherapy);
* Pregnant (if a female is of childbearing potential - defined as a pre-menopausal female capable of becoming pregnant - confirmation of pregnancy status per the site's standard of practice should be done prior to MRI);
* Unwilling or not suitable to undergo MRI or use the contrast agent gadolinium.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2018-11 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Apparent Diffusion Coefficient (ADC) | 1 year
  Whether the Apparent Diffusion Coefficient (ADC), when used systematically in conjunction with conventional Dynamic Contrast Enhanced-Magnetic Resonance Imaging (DCE-MRI), can reduce the biopsy rate by at least 20% while maintaining sensitivity.

SECONDARY OUTCOMES:
Optimal ADC Cutoffs by Lesion Type | 1 year
  Whether optimal ADC cutoffs are different for mass and non-mass lesion types;
Local and Central Review Comparison (ADC Value Differences) | 1 year
  Whether site-generated ADC values differ significantly from those obtained by central review;
Minimum B-Value for Differentiating Lesions | 1 year
  Whether the use of a nonzero minimum b-value to reduce perfusion effects in ADC calculation can increase the area under the curve (AUC) for differentiating benign and malignant lesions;
ADC Measurements/Ratios to Define Subject Lesion Variations | 1 year
  Whether the use of a normalized ADC measure (tumor/normal ratio) to account for inter- and intra-subject variations in water content and other factors can increase the AUC for differentiating benign and malignant lesions;
Combination Variables (ADC Nonzero Minimum B-Value and/or Normalized ADC) | 1 year
  Whether ADC with nonzero minimum b-value and/or normalized ADC can reduce the biopsy rate while maintaining sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Savannah Partridge, PhD, Principal Investigator — University of Washington; Habib Rahbar, MD, Study Chair — University of Washington; Thomas Chenevert, PhD, Study Chair — University of Michigan
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
see ACRIN data sharing policy : https://www.acrin.org/RESEARCHERS/POLICIES/DATAANDIMAGESHARINGPOLICY.aspx

REFERENCES:
- [Derived] McDonald ES, Romanoff J, Rahbar H, Kitsch AE, Harvey SM, Whisenant JG, Yankeelov TE, Moy L, DeMartini WB, Dogan BE, Yang WT, Wang LC, Joe BN, Wilmes LJ, Hylton NM, Oh KY, Tudorica LA, Neal CH, Malyarenko DI, Comstock CE, Schnall MD, Chenevert TL, Partridge SC. Mean Apparent Diffusion Coefficient Is a Sufficient Conventional Diffusion-weighted MRI Metric to Improve Breast MRI Diagnostic Performance: Results from the ECOG-ACRIN Cancer Research Group A6702 Diffusion Imaging Trial. Radiology. 2021 Jan;298(1):60-70. doi: 10.1148/radiol.2020202465. Epub 2020 Nov 17. PMID 33201788